CLINICAL TRIAL: NCT03992027
Title: Preventing Depression and Anxiety: A Randomized Controlled Trial of a CF-Specific CBT Intervention
Brief Title: Preventing Depression and Anxiety: A Cystic Fibrosis-Specific Cognitive Behavioral Therapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); DeltaQuest Foundation, Inc. (Unknown); University at Buffalo (Other); University of Kansas Medical Center (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Deborah Friedman, Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015P002098; FRIEDM18A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation Therapeutics, Inc)
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety
Keywords: cystic fibrosis; cognitive-behavioral therapy; prevention; coping
MeSH Terms: conditions — Depression; Anxiety Disorders; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate CF-CBT Intervention (Experimental): This group will enter immediately into the 8-session cystic fibrosis-specific cognitive-behavioral intervention program (CF-CBT).
  Interventions: Behavioral: CF-CBT: A Cognitive-Behavioral Skills-Based Program to Promote Emotional Well-Being for Adults wtih Cystic Fibrosis
- Waitlist control (Other): This group will enter into the same 8-session cystic fibrosis-specific cognitive-behavioral intervention program (CF-CBT) 3 months after enrollment.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: CF-CBT: A Cognitive-Behavioral Skills-Based Program to Promote Emotional Well-Being for Adults wtih Cystic Fibrosis — CF-CBT is an 8-session program introducing cognitive-behavioral coping skills for managing stress, and for prevention and treatment of anxiety and depression. The content of the program was developed to address stressors related to coping with cystic fibrosis. Participants will receive a patient workbook, and meet with a trained member of the CF team (interventionist) who will guide them through learning and practicing coping skills during 8 weekly sessions.
  Arms: Immediate CF-CBT Intervention
Behavioral: Waitlist Control — Participants receive usual care for 3 months followed by CF-CBT. CF-CBT is an 8-session program introducing cognitive-behavioral coping skills for managing stress, and for prevention and treatment of anxiety and depression. The content of the program was developed to address stressors related to coping with cystic fibrosis. Participants will receive a patient workbook, and meet with a trained member of the CF team (interventionist) who will guide them through learning and practicing coping skills during 8 weekly sessions.
  Arms: Waitlist control

SUMMARY:
Individuals with Cystic Fibrosis (CF) are at high risk for depression and anxiety, with negative consequences for quality of life, ability to carry out daily CF treatments, and health. CF Foundation and European CF Society guidelines recommend routine screening, treatment, and preventative efforts for depression and anxiety. Cognitive-behavioral therapy (CBT) interventions focused on teaching coping skills have a large evidence-base for prevention and treatment of depression and anxiety, but there are barriers to accessing these interventions for individuals with CF. Drs. Friedman and Georgiopoulos at Massachusetts General Hospital (MGH) have developed a CF-specific CBT-based preventive intervention for depression and anxiety with input from adults with CF and CF healthcare team members, called CF-CBT: A cognitive-behavioral skills-based program to promote emotional well-being for adults with CF, along with a training and supervision program for CF team interventionists. CF-CBT consists of 8 45-minute modules that can be flexibly delivered in the outpatient CF clinic, on the inpatient unit, or by telephone, by multidisciplinary members of the CF care team, minimizing additional cost and burden of care to patients. The goal of this study is to test CF-CBT in 60 adults screening in the mild range on measures of depression and anxiety at 4 CF centers, in a prospective randomized clinical trial comparing the intervention to usual treatment. Participants will be randomized to receive the CF-CBT intervention immediately, or to a 3-month waitlist control followed by intervention. The study will measure depression, anxiety, quality of life, stress, and coping self-efficacy before and after the CF-CBT intervention, and also 3 and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CF
* depression and anxiety scores on the PHQ-9 and/or GAD-7 screening measures in the mild but not moderate or severe range (scores are > 4 and ≤ 9)
* Able to speak and read English

Exclusion Criteria:

* Presenting an acute safety risk to self or others despite self-reporting of mild (subclinical) depression or anxiety scores on routine screening at baseline. Those reporting suicidal intent with or without specific plan will be excluded from the study. These individuals will be referred for urgent/emergent further assessment and treatment as clinically indicated.
* Participation in concomitant formal cognitive-behavioral therapy at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9) | 3 months (Baseline to Pre-intervention) for the waitlist control group; immediately post-intervention (2 to 3 months from pre-CBT assessment) for both arms; 3 months and 6 months post-intervention for both arms
  The PHQ-9 consists of nine questions measuring frequency of depressive symptoms, rated on a Likert scale from 0 "not at all" to 3 "nearly every day," with total score ranging 0-27. Clinical severity scores have been established with scores of 5, 10, 15, and 20 representing cut-off scores for mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline in Anxiety symptoms measured by the Generalized Anxiety Disorder-7 item scale (GAD-7) | 3 months (Baseline to Pre-intervention) for the waitlist control group; immediately post-intervention (2 to 3 months from pre-CBT assessment) for both arms; 3 months and 6 months post-intervention for both arms
  The GAD-7 is a 7-item measure of symptoms of anxiety. Likert scale ratings allow total scores of 0-21. Scores of 5, 10, and 15 correspond to severity ratings of mild, moderate and severe anxiety.

SECONDARY OUTCOMES:
Treatment acceptability as measured by item and total score summation on the Client Satisfaction Questionnaire (CSQ-8) with additional study-specific items | Immediately post-intervention
  The Client Satisfaction Questionnaire (CSQ-8) is an 8-item self-report measure that assesses patient service satisfaction,rated on a 4-point scale from 1=lowest to 4=highest satisfaction. Post-intervention treatment satisfaction will also be assessed with a series of structured and open-ended questions specific to the study intervention. Assessed one time immediately post-intervention.
Change from baseline in Perceived Stress measured by the Perceived Stress Scale (PSS) | 3 months (Baseline to Pre-intervention) for the waitlist control group; immediately post-intervention (2 to 3 months from pre-CBT assessment) for both arms; 3 months and 6 months post-intervention for both arms
  The PSS is a 10-item measure assessing the degree to which individuals perceive that current demands exceed their abilities to cope
Change from baseline in Cystic Fibrosis Health-Related Quality of Life measured by the adult/teen version of the Cystic Fibrosis Questionnaire-Revised (CFQ-R). | 3 months (Baseline to Pre-intervention) for the waitlist control group; immediately post-intervention (2 to 3 months from pre-CBT assessment) for both arms; 3 months and 6 months post-intervention for both arms
  The CFQ-R is a well-established measure of health-related quality of life (HrQoL). The CFQ-R contains 12 subscales, with five scales measuring physical HrQoL (Physical Functioning - 8 items; Eating Disturbances -3 items; Vitality -4 items; Respiratory - 6 items; Digestion -3 items) and seven measuring psychosocial HrQoL (e.g, Health Perceptions -3 items, Treatment Burden -3 items; Emotional Functioning - 5 items; Social Functioning -6 items; Body Image -3 items; Role Functioning - 4-items). Items are rated on 4-point Likert scale with higher scores reflecting better quality of life. Scaled scores are obtained for each subscale.
Change from baseline in Coping Self-Efficacy measured by the CF Coping Self-Efficacy Measure developed for this study | 3 months (Baseline to Pre-intervention) for the waitlist control group; immediately post-intervention (2 to 3 months from pre-CBT assessment) for both arms; 3 months and 6 months post-intervention for both arms
  The CF Coping Self-Efficacy measure includes 25 items and was developed for this study to assess patient-reported confidence in their ability to use CBT coping skills that are introduced in the CF-CBT intervention to manage general stressors and those related to having CF. Each item is rated on a 10-point Likert scale from 10 to 100 from "very uncertain" to "very certain" about the ability to use each skill , with higher scores indicating greater confidence in being able to use coping skills. Mean scores are obtained for each of 5 proposed subscales (Relaxation; Behavioral Activation; Adaptive Thinking/Cognitive Restructuring; Active Coping/Problem-Solving; and CF-Specific Coping).
Feasibility of the intervention will be indicated by Rate of Attrition, or rate of drop-out or non-completion of the CF-CBT program once enrolled | From baseline to post-intervention (2 to 3 months for the immediate intervention arm; 5 to 6 months for the waitlist arm)
  Rate of attrition will be summarized by calculating the percentage of CF-CBT sessions completed by participants over the course of the study period. The CF-CBT program consists of 8 sessions, and the proposed sample size of the study will be 60 participants, such that an Attrition Rate of 0% would be calculated if all 480 CF-CBT sessions were completed.
Feasibility of the intervention will also be indicated by Treatment Fidelity, measured as percent adherence to general and CF-CBT session-specific objectives. | 2 years and 3 months (Over the course of the study period)
  Treatment Fidelity will be rated independently for a random 20% of CF-CBT sessions. Each session that is rated will have a general objectives and session-specific objectives rating. The general objectives rating includes 6 items rated on a 6-point Likert scale from "poor/not at all" to "Excellent," with total score ranging from 0-36. Session-specific objectives will include between 5 and 7 items that are dichotomous indicating whether or not (yes/no) a specific objective was met. A percentage of the possible total will be calculated for both general and session-specific objectives for each rated session. All CF-CBT sessions will be recorded so that a random 20% may be independently rated. The initial 8 sessions for each newly trained interventionist will be excluded from analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Friedman, PhD, Principal Investigator — Massachusetts General Hospital; Anna Georgiopoulos, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Stanford University, Palo Alto, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No